CLINICAL TRIAL: NCT02285361
Title: A Regulatory Requirement Post-marketing Surveillance Study to Monitor the Safety and Efficacy of GIOTRIF® (Afatinib Dimaleate, 20mg, 30mg, 40mg, q.d) in Korean Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) With Epidermal Growth Factor Receptor (EGFR) Mutations or Patients With Locally Advanced or Metastatic NSCLC of Squamous Histology Progressing on or After Platinum-based Chemotherapy
Brief Title: GIOTRIF rPMS in Korean Patients With NSCLC
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200.235
Record Dates: First submitted 2014-10-20; First posted 2014-11-07 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- GIOTRIF
  Interventions: Drug: GIOTRIF 20mg; Drug: GIOTRIF 40mg; Drug: GIOTRIF 30mg

INTERVENTIONS:
Drug: GIOTRIF 20mg — NSCLC with GIOTRIF 20mg
Drug: GIOTRIF 40mg — NSCLC with GIOTRIF 40mg
Drug: GIOTRIF 30mg — NSCLC with GIOTRIF 30mg

SUMMARY:
To monitor the safety profile and efficacy of GIOTRIF® (afatinib dimaleate, q.d) in Korean patients with locally advanced or metastatic non-small cell lung cancer (NSCLC)

ELIGIBILITY:
Inclusion criteria:

1. Patients who have been started on GIOTRIF® in accordance with the approved label in Korea
2. Age = 19 years at enrolment
3. Patients who have signed on the data release consent form

Exclusion criteria:

1. Known hypersensitivity to afatinib or any of its excipients
2. Patients with rare hereditary conditions of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
3. Patients for whom GIOTRIF® is contraindicated according to the local label

Ages: 19 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC in Korea
Sampling Method: Probability Sample
Enrollment: 1272 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, South Korea

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an observational prospective, non-interventional, open-label, multi-centre national study in Korean patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) with Epidermal Growth Factor Receptor (EGFR) mutations or patients with locally advanced or metastatic NSCLC of squamous histology progressing on or after platinum-based chemotherapy
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- GIOTRIF®: GIOTRIF® was prescribed according to the local label and at the discretion of the treating physician. The physicians indicated doses and timing based on the current authorized label in Korea. Possible dosage were 20 milligram (mg), 30 mg and 40 mg administered orally, once daily, at least 1 hour before a meal or at least 3 hours after a meal, taken without food and swallowed whole with water.
Period: Overall Study
Arm/Group | GIOTRIF®
Started | 1272
Completed (All Participants whose case report forms (CRFs) were retrieved during the re-examination period and who did not violate the inclusion/exclusion criteria.) | 1221
Not Completed | 51
Not completed — Protocol Violation | 43
Not completed — Lost to Follow-up | 5
Not completed — Not taken GIOTRIF | 2
Not completed — Consented prior to the contract date | 1

BASELINE CHARACTERISTICS:
Population: All Participants whose case report forms (CRFs) were retrieved during the re-examination period (29 Jan 2014 - 28 Jan 2020) and who did not violate the inclusion/exclusion criteria. 1 subject was excluded from the set based on disease indication.
Arm/Group | GIOTRIF®
Number analyzed (Participants) | 1220
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.26 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 662
  Male | 558
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs)
Description: Percentage of participants with Adverse Drug Reactions (ADRs).
Time Frame: From baseline (Visit 1) until last visit (the last follow-up visit a patient actually attended during the study), up to 1051 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | GIOTRIF®
Number analyzed (Participants) | 1220
Percentage of participants | 89.92

2. Secondary Outcome: Progression-Free Survival (PFS) Rate at 48 Weeks
Description: Progression-Free Survival (PFS) rate, defined as the percentage of patients who were alive and without disease progression at the 48-week tumour assessment. Progression was assessed by the investigator according to local standard pattern of care for non-small cell lung cancer (NSCLC).
  If a patient is known to have progressed, but the date of progression is not attainable, the last date when the patient was assessed will be used as date of progression.
  PFS rate at 48 weeks was estimated using Kaplan-Meier estimates on the PFS curve.
Time Frame: From week 0 until week 48. Up to 48 weeks.
Population: Effectiveness assessment set: all participants whose case report forms (CRFs) were retrieved during the re-examination period (29 Jan 2014 - 28 Jan 2020) and who did not violate the inclusion/exclusion criteria. 221 subjects were excluded due to missing effectiveness assessments.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GIOTRIF®
Number analyzed (Participants) | 1000
Percentage of participants | 73.74 [70.37 to 76.80]

3. Secondary Outcome: Percentage of Participants With Best Response
Description: Best response is defined as the best response observed in individual subject from the date of the first administration of the study medication until the earliest recording of Progressive disease (PD), death, or end of treatment (as long as no additional anti-cancer therapy was implemented). Disease Assessment will be based on the assessment of cancer related symptoms and, if available, radiologic assessments as per standard of care at the site.
  Tumour response according to investigator's assessment
  Each patient will be assigned to one of the following categories:
  1. Complete response (CR)
  2. Partial response (PR)
  3. Stable disease (SD)
  4. Progressive disease (PD)
  5. Not evaluable for response, reasons to be specified (e.g. early death, tumour assessments incomplete, etc.)
Time Frame: Tumour assessments performed at week 0, 8±2, 24±2 and 48±2. Up to 50 weeks.
Population: Effectiveness assessment set: all participants whose case report forms (CRFs) were retrieved during the re-examination period (29 Jan 2014 - 28 Jan 2020) and who did not violate the inclusion/exclusion criteria. 221 subjects were excluded due to missing effectiveness assessments, an additional 36 subjects were excluded for not completing the assessment at the last visit.
Measure: Number; unit: Percentage of participants
Arm/Group | GIOTRIF®
Number analyzed (Participants) | 964
Percentage of participants
  Complete Response | 2.90
  Partial Response | 60.89
  Stable Disease | 32.26
  Progressive Disease | 3.22
  Not Evaluable | 0.73

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS), defined as time from the date of the first administration of afatinib to the date of death. Kaplan-Meier estimates and 95% confidence intervals for the 25th, median, and 75th percentiles of the survival distribution will be calculated for OS.
  For patients with known date of death:
  OS [days] = date of death - (date of start of treatment) + 1
  For patients known not death case:
  OS (censored) [days] = date of last contact showing no death - (date of start of treatment) + 1.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | GIOTRIF®
Number analyzed (Participants) | 1000
Days | NA [1051 to NA] — The median and upper confidence interval could not be estimated due to the low number of deaths.

ADVERSE EVENTS:
Time Frame: From baseline (Visit 1) until last visit (the last follow-up visit a patient actually attended during the study), up to 1051 days.
Description: For this non interventional study, all 1272 participants whose case report forms (CRFs) were retrieved during the re-examination period (29 Jan 2014 - 28 Jan 2020) and who did not violate the inclusion/exclusion criteria were included. Among these, 6 participants were deemed not eligible retrospectively and were additionally excluded.
Arm/Group | GIOTRIF®
All-Cause Mortality (participants affected / at risk) | 52/1266
Serious Adverse Events (participants affected / at risk) | 442/1266
Other Adverse Events (participants affected / at risk) | 1076/1266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GIOTRIF® (N=1266)
Anaemia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 4
Otolithiasis (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Thyroid mass (Endocrine disorders) | 1
Glaucoma (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 53
Dysphagia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 11
Chest pain (General disorders) | 1
Death (General disorders) | 4
Disease progression (General disorders) | 99
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Pyrexia (General disorders) | 4
Cholelithiasis (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Atypical pneumonia (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chest wall abscess (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Eczema herpeticum (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Infectious pleural effusion (Infections and infestations) | 1
Onychomycosis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 35
Pneumonia bacterial (Infections and infestations) | 2
Pneumonia viral (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 2
Renal abscess (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Subcutaneous abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Compression fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2
Meniscus injury (Injury, poisoning and procedural complications) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Liver function test increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 4
Lactic acidosis (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 100
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 4
Embolic cerebral infarction (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Hemiparesis (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Myelopathy (Nervous system disorders) | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 4
Disorientation (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 19
Azotaemia (Renal and urinary disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 22
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Hypovolaemic shock (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Pelvic venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GIOTRIF® (N=1266)
Diarrhoea (Gastrointestinal disorders) | 866
Nausea (Gastrointestinal disorders) | 91
Stomatitis (Gastrointestinal disorders) | 377
Paronychia (Infections and infestations) | 314
Decreased appetite (Metabolism and nutrition disorders) | 204
Pruritus (Skin and subcutaneous tissue disorders) | 166
Rash (Skin and subcutaneous tissue disorders) | 515

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT02285361/Prot_SAP_000.pdf